CLINICAL TRIAL: NCT03785665
Title: To Monitor the Whole Gut Transit Time and Repeatability of the Motility of MD1 Capsules in the Colon of Subjects With Known Polyps and in Healthy Subjects
Brief Title: Motility of the Check-cap's MD1 Colon Capsule in Subjects Following Colon Rectal Cancer Screening by Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-MD1-01-0097
Record Dates: First submitted 2018-11-28; First posted 2018-12-24 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Multi-Center, Open, Home Monitoring, Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): All study participants will be examined by the MD1 capsules, 2-5 capsules per person, one capsule at a time. Efforts will be made to maintain balanced numbers between men and women and even distribution of ages
  Interventions: Device: MDI

INTERVENTIONS:
Device: MDI — Capsule MD1 (Motility dummy 1)
  Other Names: Capsule MD1 (Motility dummy 1)

SUMMARY:
To monitor the Whole Gut Transit Time and repeatability of the motility of MD1 capsules in the colon of subjects with known polyps and in healthy subjects. Multi-Center, Open, Home Monitoring, Prospective Study. Up to 100 participants in various phases 2-5 capsules per person, (1 capsule at a time) The primary objective of the study is to monitor the variability of the motility of the MD1 capsules in the Gastrointestinal tract of human subjects with and without polyps in previous Colonoscopy.

DETAILED DESCRIPTION:
The subject population in this study will be composed of male and female subjects older than 40 and younger than 80 years old who volunteer for the experiment and qualify with the inclusion / exclusion criteria A total of one hundred (100) subjects will be enrolled in this study. All study participants will be examined by the MD1 capsules, 2-5 capsules per person, one capsule at a time. Efforts will be made to maintain balanced numbers between men and women and even distribution of ages.

The study will be conducted by phases:

A 15-20 Men with polyps in previous Colonoscopy (2-3 repeated ingestions) B. 10-20 Men With no polyps in previous Colonoscopy (1-2 repeated ingestions) C. 15-20 Women with polyps in previous Colonoscopy (2-3 repeated ingestions) D. 10-20 Women With no polyps in previous Colonoscopy (1-2 repeated ingestions) E Same as A-D with the use of prokinetic drugs F. Same as A-D with different type of capsules (lower weight and/or rounded caps on both sides).

The total duration of the study for each subject is two-four weeks. Each subject will ingest 2-5 capsules, one at a time, with at least 1 week apart between repeated ingestion

1. st Visit (phone interview) - Each subject will receive a comprehensive explanation regarding the study nature. During this process, and per ethical committee approval, subjects may be asked several questions (over the phone) regarding their medical background for preliminary assessment of eligibility.
2. nd Visit - Once informed consent is obtained, a thorough evaluation of subject's eligibility will be performed based on inclusion / exclusion criteria.

Consent to participate in this study must be given in writing. The signed informed consent will remain in subject's file. A signed copy will be given to the subject.

Subject will ingest the capsule (in the presence of a medical professional).

Post ingestion, the subject will receive detailed instructions about the daily routine and activities and then will be discharged home with written instructions on the procedure (IFU - Instructions for use). The subject should avoid intensive physical exercise during the procedure or any extreme activities. The subject should make an effort to stay at home or other familiar surroundings (within 2 hours of driving from the clinic), and may continue daily activities such mobile/computer/TV (Television) use, shower, sleep or eat.

Details on allowed and restricted activities are listed in the Information For use which is included in the Kit).

All subjects will be provided with a contact card with study details and site contact information (24/7).

Discharged home

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 40 and 80 years of age
* Subjects which are generally healthy
* Subjects who were examined by colonoscopy during the previous 5 years period and can provide a copy of the report
* Subjects who are ready to undergo the monitoring routine and commit to at least two experiments
* Signed informed consent.

Exclusion Criteria:

* Subjects with advanced cancer or other life threatening diseases or conditions
* Subject with known history of dysphagia or other swallowing disorders
* Subject with known history of Gastrointestinal disease or symptoms, such as: Crohn's disease, Colitis, Inflammatory bowel disease (IBD), Meckel's Diverticulum, Bowen Hernia, Mega Colon, fistulas or other strictures (doctors' discretion).
* Subject with known motility disorder or Chronic Constipation (less than 3 bowel movements/week)
* Subject with known delayed gastric emptying
* Subject with prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by physician discretion
* Subject with any condition believed to have an increased risk for capsule retention such as intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or Nonsteroidal anti-inflammatory drugs (NSAID) enteropathy, as determined by physician discretion
* Subjects with known sensitivity to iodine, or with kidney failure
* Subjects with morbid obesity (Body Mass Index > 35)
* Subjects with belly / girth circumference > 125 cm
* Subject with any known condition which precludes compliance with study and/or device instructions
* Subject with known condition of drug abuse and/or alcoholism
* Women who are either pregnant or nursing at the time of screening (to be verified by test in case of woman of child-bearing potential that do not practice medically acceptable methods of contraception)
* Concurrent participation in another clinical trial using any investigational drug or device

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Measure the variability of the motility (Whole gut transit time from ingestion to excretion {hours}) of the MD1 (Motility dummy 1) capsules in the Gastrointestinal tract of human subjects with and w/out polyps in previous Colonoscopy. | 12 months
  All participating subjects will be consented for multiple measurements. In selected subjects the experiment will be repeated with same type MD1 capsule but w/out the drug, to compare the effect of the drug on the motility and the instantaneous speed during contractions. These subjects will be selected according to their results in the first round, ease of adjustment to the monitoring routine, retrieval of the excreted capsules and lack of any side effects or complains.
  The repeated procedure will be at least 1 week apart and will be approved by the investigator only after positive identification of the excretion of the first capsule. Naturally, there is no need to repeat the colonoscopy procedure The repeated tests will be conducted according to the same protocol. There are no additional safety issues in the re-ingestions tests since the 1st capsule has to be excreted and retrieved few days before the repeated experiment starts

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Shpigelman, Study Director — VP R&D
Locations (1):
- Bnai Zion Medical Center, Haifa, North, Israel